CLINICAL TRIAL: NCT06364046
Title: Efficacy and Safety of DEB-BACE Combined With Serplulimab in First-line Treatment of SCLC:A Prospective, Single-center, Randomized, Open, Double-arm Clinical Trial
Brief Title: Efficacy and Safety of DEB-BACE Combined With Serplulimab in First-line Treatment of SCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJLS-KLDMIR-22006
Record Dates: First submitted 2024-03-14; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma; Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Programmed Cell Death Protein 1 Inhibitor; Serplulimab; Drug-eluting beads bronchial arterial chemoembolization
MeSH Terms: conditions — Carcinoma; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting Beads Bronchial Arterial Chemoembolization Combined with Serplulimab (Experimental)
  Interventions: Procedure: Drug-eluting beads bronchial arterial chemoembolization; Drug: Serplulimab
- Irinotecan Single-agent Intravenous Chemotherapy Combined with Serplulimab (Active Comparator)
  Interventions: Drug: Serplulimab; Procedure: Intravenous chemotherapy

INTERVENTIONS:
Procedure: Drug-eluting beads bronchial arterial chemoembolization — Drug-eluting beads bronchial arterial chemoembolization generally uses platinum-containing two-drug chemotherapy "platinum (cisplatin, carboplatin, nedaplatin) combined treatment, and drug-loaded microspheres are loaded with irinotecan. The dose of chemotherapy drugs is set to 75mg/m2 of platinum, and the dose of chemotherapy through catheter infusion is reduced by 25%. The dose of drug-loaded drugs is irinotecan 80mg/ m2. Chemotherapy was perfused first, followed by embolization with drug-loaded microspheres, until the blood flow in the artery supplying the tumor slowed down and approached stagnation. The number of DEB-BACE treatments is determined by the investigator, and is given as needed according to the patient's condition, usually 1-2 times, with an interval of 28±10 days.
  Arms: Drug-eluting Beads Bronchial Arterial Chemoembolization Combined with Serplulimab
Drug: Serplulimab — Programmed cell death protein 1 inhibitor fixation was treated with serplulimab (Fuhong Hanlin Co., LTD.). It is administered by intravenous infusion, and the recommended dose is 200 mg, given once every 21 days. The medication will last for two years until disease progression or intolerable toxicity occurs. During immunotherapy, immunosuppressive agents will not be replaced and the dose will not be adjusted.
Procedure: Intravenous chemotherapy — Intravenous chemotherapy with irinotecan 65mg/m2 on day 1 and day 8, given once every 21 days
  Arms: Irinotecan Single-agent Intravenous Chemotherapy Combined with Serplulimab

SUMMARY:
This project aims to conduct a prospective, single-center, randomized, open-label, two-arm study to compare the clinical efficacy and safety of bronchial arterial chemoembolization with drug-eluting beads (DEB-BACE) combined with serplulimab versus conventional intravenous chemotherapy combined with Serplulimab as first-line treatment for SCLC patients. The objective is to provide evidence-based support for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old, regardless of gender;
* SCLC diagnosis based on histopathology according to the Primary Lung Cancer Diagnosis and Treatment Guidelines (2018 edition);
* TNM stage II-IV;
* ECOG PS score ≤2;
* Predicted survival time more than 3 months;
* Provision of signed informed consent.

Exclusion Criteria:

* Previous interventional therapies such as iodine seed implantation (within the past six months), ablation, BACE, or immunotherapy;
* Concurrent presence of other incurable malignant tumors;
* White blood cell count less than 3×10^9/L, neutrophil absolute count less than 1.5×10^9/L, neutrophil/lymphocyte ratio equal to or greater than 3, platelet count less than 50×10^9/L, hemoglobin concentration less than 90 g/L;
* Hepatic and renal insufficiency (creatinine level exceeding 176.8μmol/L); Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels more than twice the upper limit of normal;
* Uncorrectable coagulopathy or concurrent active hemoptysis;
* Complicated with active infection requiring antibiotic treatment;
* Uncontrolled hypertension, diabetes, or cardiovascular disease;
* Allergy to contrast agents;
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Proportion of patients who achieved complete remission (CR) or partial remission (PR) according to mRECIST criteria at 1 month, 3 months, and 6 months , assessed up to 12 months
  Evaluation index of clinical efficacy of anticancer drugs.

SECONDARY OUTCOMES:
Progression Free Survival | The time from enrollment to tumor progression or death from any cause, whichever came first, measured in "months", assessed up to 2 years
  The most common primary endpoint in cancer trials.
Overall Survival | Time from randomization to death from any cause, in "months", assessed up to 2 years. For patients who are still alive at the time of data analysis, OS is calculated based on the date when the patient is last known to be alive.
  The best efficacy endpoint in cancer clinical trials.
Time to tumor untreatable progression | The time interval between randomization to tumor progression that patients are unable to further receive treatment, assessed up to 12 months.
  End point of antitumor drug trial.
Disease Control Rate | Proportion of patients with complete remission (CR), partial remission (PR), and stable disease (SD) according to mRECIST criteria, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs
Duration of Overall Response | The time from the first assessment of the tumor as complete remission or partial remission to the first assessment as disease progression or death from any cause, assessed up to 12 months
  Evaluation index of clinical efficacy of anticancer drugs.
Tumor biomarkers | From pre-procedure to every follow-up time, assessed up to 2 years.
  carcinoembryonic antigen, carbohydrate antigen 125, squamous cell carcinoma, etc
Tumor biomarkers | From pre-procedure to every follow-up time, assessed up to 2 years.
  squamous cell carcinoma
Tumor biomarkers | From pre-procedure to every follow-up time, assessed up to 2 years.
  carbohydrate antigen 125
Tumor biomarkers | From pre-procedure to every follow-up time, assessed up to 2 years.
  carcinoembryonic antigen
Eastern Cooperative Oncology Group Score | The patient's performance status score is divided into 6 grades. The lowest grade is 0, and the highest grade is 5. The patient's physical state deteriorates as the grade rises,assessed up to 2 years..
  Time Frame: From pre-procedure to every follow-up time, assessed up to 2 years.
Recurrence rate of hemoptysis | From date of randomization to every follow-up time, assessed up to 2 years.
  Hemoptysis occurs again
Quality of life Questionare-Core score | From date of randomization to every follow-up time, assessed up to 2 years.
  The European Organization for Reasearch and Treatment of Cancer Quality of life Questionare-Core score. All items and subscales were converted from 0 to 100, with higher scores indicating better overall quality of life.
The incidence of adverse events and serious adverse events | Time Frame: From date of randomization to every follow-up time, assessed up to 2 years.
  Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Pain assessment | From date of randomization to every follow-up time, assessed up to 2 years.
  Visual Analogue Scale/Score.The tool is a 10 cm long roving ruler with 11 scales ranging from 0 to 10. A score of 0 means no pain, and a score of 10 means unbearable pain. The higher the score, the more severe the pain

CONTACTS AND LOCATIONS:
Overall Officials: Linqiang Lai, MD., Study Director — The Central Hospital of Lishui City
Locations (1):
- Lishui central hospital, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers.
  Shared data does not provide any private information of the participants.